CLINICAL TRIAL: NCT04591145
Title: Validation of a Deep Learning Based Bowel Preparation Evaluation System: A Prospective, Multi-center, Cross-sectional Study
Brief Title: Multi-center Validation of a Deep Learning Based Bowel Preparation Evaluation System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan Central Hospital (Other); Wuhan Third Hospital (Other); The General Hospital of Central Theater Command (Other); The Third People's Hospital of Hubei Province (Other); Wuhan Puren Hospital (Other); Wuhan Puai Hospital (Unknown); Tian You Hospital Affiliated to Wuhan University of Science and Technology (Unknown); Wuhan Red Cross Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: EA-20-002
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Adenoma; Bowel Preparation
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients received bowel preparation and colonoscopy. The withdrawal phase video was saved and their lesions detection was record.
  Interventions: Other: Observational group

INTERVENTIONS:
Other: Observational group — Patient receive the standard bowel preparation strategy and routine colonoscopy

SUMMARY:
A deep learning based system to calculate the proportion of Boston Bowel Prep Scale (BBPS) score of 0-1 during withdrawal phase has been constructed previously. This multi-center study is going to perform a prospective observational study to validate the threshold of the adequate proportion.

DETAILED DESCRIPTION:
Inadequate bowel preparation is insufficient for identification of polyps greater than 5 mm. However, bowel preparation assessment involved subjectivity and uncertainty. We constructed a deep learning based system to calculate the proportion of Boston Bowel Prep Scale (BBPS) score of 0-1 during withdrawal phase and performed a prospective observational study to validate the threshold of the adequate proportion.The multi-center study is aimed to verify the extrapolation and robustness of the scoring threshold based on artificial intelligence intestinal cleanliness evaluation system explored in the early stage, and propose a more accurate and quantifiable threshold for evaluating the eligibility of intestinal preparation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above;
* Ability to read, understand and sign informed consent forms;
* The researchers believe that the subjects can understand the process of the clinical study and are willing and able to complete all the study procedures and follow-up visits to cooperate with the study procedures.

Exclusion Criteria:

* Patients with contraindications to colonoscopy (obstruction or perforation, severe acute inflammatory bowel disease, toxic megacolon, severe heart failure, severe heart failure, etc.);
* Patients with galactosemia;
* Pregnant or lactating women;
* Patients used lactulose, a stimulant, or laxative within 7 days;
* Patients refused to sign informed consent forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Continuous colonoscopy from October to December 2020 will be collected in our participating general hospitals.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2020-10-09 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cleanliness assessment of different intestinal segment in the artificial intelligence system | 3 Months
  The Artificial intelligence evaluates the Boston Bowel Preparation score of the ascending colon, transverse colon and descending colon in real-time, and calculates the proportion of 0-1 Score
Adenoma detection rate | 3 Months
  The numerator is the number of cases of adenomas detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.

SECONDARY OUTCOMES:
Advanced adenoma detection rate | 3 Months
  The numerator is the number of cases of advanced adenomas detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.
Polyps detection rate | 3 Months
  The numerator is the number of cases of polyps detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.
The mean number of adenomas per procedure | 3 Months
  The numerator is the total number of polyps detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy
Detection rate of large, small and diminutive polyps | 3 Months
  The numerator was the number of patients with large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
The mean number of large, small and diminutive polyps per procedure | 3 Months
  The numerator was the number of large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of large, small and diminutive adenomas | 3 Months
  The numerator was the number of patients with large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
The mean number of large, small and diminutive adenomas per procedure | 3 Months
  The numerator was the number of large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of adenoma in different sites | 3 Months
  The numerator is the number of cases of adenoma detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
The mean number of adenomas in different sites per procedure | 3 Months
  The numerator is the total number of adenomas detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Time of colonoscopic insertion/withdrawal | 3 Months
  The duration of colonoscopic insertion from rectum to ileocecal valve or appendiceal opening and the duration of colonoscopic withdrawal from ileocecal valve or appendiceal opening to colonoscopy finished.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China